CLINICAL TRIAL: NCT06500728
Title: Visual Involvement in Giant Cell Arteritis
Acronym: Visu-GCA
Status: Recruiting | Type: Observational
Sponsor: ASST Fatebenefratelli Sacco (Other)
Responsible Party: Principal Investigator, Enrico Tombetti, Co-Principal Investigator, ASST Fatebenefratelli Sacco
Other Study IDs: Visu-GCA Trial
Record Dates: First submitted 2024-07-07; First posted 2024-07-15 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Giant Cell Arteritis; Visual Impairment; Central Retinal Artery Occlusion; Anterior Ischemic Optic Neuropathy; Paracentral Acute Middle Maculopathy; Posterior Ischemic Optic Neuropathy; Retinal Ischemia; Blindness; Visual Disorder
Keywords: Giant Cell Arteritis; Visual impairment; Optical Coherence Tomography (OCT); High resolution Optical Coherence Tomography (HR-OCT); Angio-Optical Coherence Tomography (OCT-A); Fluorescein angiography; Indocyanine green angiography
MeSH Terms: conditions — Giant Cell Arteritis; Vision Disorders; Retinal Artery Occlusion; Optic Neuropathy, Ischemic; Blindness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- GCA patients: Patients older than 18 years with clinically suspected or confirmed giant cell arteritis, who experience newly diagnosed visual impairment with suspected or confirmed correlation with vasculitis.
  Interventions: Diagnostic Test: Fluorescein and Indocyanine green Angiography; Diagnostic Test: High-resolution Optical Coherence Tomography; Diagnostic Test: Angio-Optical Coherence Tomography
- Non arteritis patients: Patients over 18 years of age who experience newly diagnosed acute visual impairment with GCA phenotypes (e.g. AION, CRAO) but without any correlation with vasculitis aetiology.
  Interventions: Diagnostic Test: Fluorescein and Indocyanine green Angiography; Diagnostic Test: High-resolution Optical Coherence Tomography; Diagnostic Test: Angio-Optical Coherence Tomography

INTERVENTIONS:
Diagnostic Test: Fluorescein and Indocyanine green Angiography — The ophthalmologist frequently recommends fluorescein (FAG) and indocyanine green angiography (ICGA) at baseline (T0) to evaluate retinal and choroidal vascularisation. They can be repeated also after 48-72 hours (T1), 7 ± 2 days (T2), 4 ± 1 weeks (T3), 12 ± 2 weeks (T4) or 26 ± 2 weeks (T5).
  Other Names: FAG and ICGA
Diagnostic Test: High-resolution Optical Coherence Tomography — The ophthalmologist often suggests performing HR-OCT initially (T0) to assess the width of the macula and optic nerve with potential signs of ischemic lesions in these areas. This assessment can also be repeated after 48-72 hours (T1), 7 ± 2 days (T2), 4 ± 1 weeks (T3), 12 ± 2 weeks (T4), or 26 ± 2 weeks (T5).
  Other Names: HR-OCT
Diagnostic Test: Angio-Optical Coherence Tomography — The ophthalmologist often suggests OCT-A at the beginning (T0) to assess the retinal and choroidal vascularization. These tests can also be done after 48-72 hours (T1), 7 ± 2 days (T2), 4 ± 1 weeks (T3), 12 ± 2 weeks (T4), or 26 ± 2 weeks (T5).
  Other Names: OCT-A

SUMMARY:
This observational study aims to enhance the description of the different ways Giant Cell Arteritis (GCA) affects vision. The latest technology and knowledge are used to improve how we diagnose and predict patient outcomes. GCA is the most frequent vasculitis, an inflammation of vessels, in older adults. It involves large and medium-sized arteries and causes ischemic alterations such as stroke and blindness, through damage of extracranial arteries.

The primary objective is to compare the frequency of the various ocular findings between the main alterations of arteritic and non-arteritic aetiology, such as Arteritic Anterior Ischemic Optic Neuropathy (A-AION) Vs. Non-Arteritic Anterior Ischemic Optic Neuropathy (NA-AION) or Central Retinal Artery Occlusion (CRAO) from GCA Vs. from other causes, through a comprehensive clinical and instrumental evaluation.

DETAILED DESCRIPTION:
Giant-cell arteritis (GCA) is an idiopathic inflammatory condition affecting medium- and large-sized arteries. This condition typically affects females over 50, with a peak incidence in the eighth decade of life. It is a rare disease, with an annual incidence in southern Europe (including Italy) of approximately 12/100000 inhabitants aged > 50 years. This clinical condition has considerable heterogeneity among patients, with different clinical phenotypes recognised, predominantly involving the large vessel (LV-GCA) and the medium-sized arteries of the cephalic district (cGCA). The main complications of cephalic involvement are ischaemic events such as stroke and optic involvement. Visual involvement is a minor but the main prognostic factor in patients with GCA, as it can lead to irreversible vision loss. Patients with visual involvement often exhibit other disease features but with a less intense inflammatory response compared to subjects without visual involvement. Ocular involvement occurs with a wide clinical spectrum of ocular manifestations, from amaurosis fugax and diplopia to permanent loss of visual capacity. This irreversible or partially reversible visual impairment is mainly linked to three mechanisms:

* Arteritic anterior ischaemic optic neuropathy (A-AION), which is present in 90% of cases of irreversible vision loss; it is secondary to ischaemic involvement of the short posterior ciliary arteries that supply the optic nerve head; direct ophthalmoscopy shows typically an oedematous and pale optic disc, with a resolution in cupping characteristics like in glaucomatous optic neuropathy after 4 weeks. In the presence of cilio-retinal artery, the vascular territory of this arterial variation could be involved. This ophthalmological image is being considered for differential diagnosis with non-arteritic anterior ischemic optic neuropathy (NA-AION). NA-AION is caused by a compartment syndrome that occurs at the level of the optic nerve head. This is triggered by even transient hypoperfusion that causes ischemic swelling in an area with little room to expand at the level of the lamina cribrosa. As the therapy is completely different, the differentiation between A-AION and NA-AION is crucial: Hayreh et al. differ these conditions according to the extra-ocular features of GCA and the ophthalmological characteristics (presence of pallor/papillary haemorrhages, cilio-retinal occlusion if arising from a territory with choroidal ischaemia and evidence of choroidal ischaemia or delayed choroidal perfusion).
* In 15% of cases, internal retinal ischaemia occurred during GCA due to involvement of the central retinal artery (CRAO) or one of its branches (BRAO). Direct ophthalmoscopy shows peripheral retinal whitening in contrast to the cherry-red macula. Sub-occlusive involvement of the retinal vasculature provides necrotic spots of certain retinal layers, providing superficial cottony exudates and deep paracentral acute middle maculopathy (PAMM). PAMM was first described in 2013. A single study about 52 patients with visual GCA observed PAMM in 26% of patients, either isolated or in association with other forms of visual involvement. However, this diagnosis requires evaluation by Optical Coherence Tomography (OCT).
* In 5% of cases of GCA, posterior ischemic optic neuropathy (PION) occurs due to altered circulation in the retrobulbar optic nerve. No typical retinal or optic nerve changes are evident on direct ophthalmoscopy.

Various unmet needs in the ophthalmological literature could impact on the management of patients with acute visual impairment in suspected GCA:

1. Semeiological aspects of the rare visual phenotypes are described in studies with sample sizes ranging between 8 and 85 subjects. Multicenter studies with the largest sample sizes and ten-year recruitment do not explain deeply all ophthalmological pictures meanwhile small studies interfere with a clear description of the entire spectrum of ophthalmic semeiotic manifestations, highlighting only the most frequent phenotypes and making diagnosis very complex to date. In this center, among 60 patients enrolled in the last 3 years, 5 patients with PAMM and 2 with atypical A-AION were described, complicating the diagnostic-therapeutic procedure.
2. Types of enrolled GCA patients are a limiting aspect, due to the evolution of vasculitis definition, diagnosis and management (i.e. last updated in American College of Rheumatology guidelines of 2022) and awareness about diagnosis delay and visual prognosis. Therefore, it is important to define ophthalmological manifestations and frequency distributions in enrolled patients according to recent criteria and current clinical practices.
3. Many studies with an ophthalmological focus were published several years ago. New ophthalmological clinical pictures have been recognised (such as PAMM, in 2013) and ophthalmology-focused instrumental technology has advanced considerably, such as high-OCT, Optical Coherence Resonance (OCR) and angio-Optical Coherence Tomography (OCT-A). Moreover, considering that extra-ocular manifestations of GCA may be absent in approximately 20% of patients with visual involvement, it is particularly important to update semeiological knowledge and predictive and prognostic values.
4. PAMM in GCA was described in a few epidemiological studies with a small sample size. Although PAMM could represent the second most frequent form of visual impairment in GCA, OCT is not yet widely used and/or practised in comparison with traditional methods such as ophthalmoscopy and fluoroangiography.

This observational study aims to improve the ophthalmological description of different visual involvement phenotypes in GCA. This will be achieved by utilizing state-of-the-art technology and nosographic knowledge to improve patient diagnosis and prognostic stratification.

The primary objective is a comparison of the frequency of the various semeiological findings by multi-parametric evaluation, among the main pathological ocular alterations of arteritic and non-arteritic aetiology (e.g. A-AION Vs. NA-AION, CRAO from arteritis Vs. CRAO from other causes). The second objectives are:

* Prevalence of the GCA visual phenotypes, including the potential co-existence of several of them (e.g. paracellular retinal ischemia as in PAMM, choroidal and papillary ischemia).
* Integration of clinical findings with ophthalmological methods such as visual acuity, campimetry, retinal fluorangiography, OCT, and OCT-A in various pathological visual conditions.
* Temporal evolution of the visual acuity and semeiological findings after therapy and correlation with prognosis.

This prospective study enrolls patients referred to the emergency room or ophthalmology outpatient clinic for new-onset visual symptoms, for which they will perform the clinical, laboratory and instrumental examinations required by existing clinical practice. For patients with suspected GCA, venous blood samples (18 ml per sample) are scheduled at baseline, and at times 7 days, 3 months and 6 months.

Clinical management and treatment will follow international recommendations per the 2021 American College of Rheumatology (ACR) and 2018 European Alliance of Associations for Rheumatology (EULAR) guidelines, due to the progression of acute visual impairment leading to permanent visual loss. Ophthalmological assessment will be scheduled at baseline (T0), which is repeated after 48-72 hours (T1), 7 ± 2 days (T2), 4 ± 1 weeks (T3), 12 ± 2 weeks (T4) and 26 ± 2 weeks (T5). At each time point, the evaluation includes an assessment of visual acuity, fundus, and visual field. The ophthalmologist frequently recommends fluorescein (FAG) and indocyanine green angiography (ICGA), OCT with high-resolution technique, and OCT-A. In addition to the ophthalmological assessment, patients will also undergo an internal and immuno-rheumatological evaluation to address the management and treatment of the underlying condition causing the visual impairment. Internal or immuno-rheumatology follow-up will depend on the underlying diagnosis and follow normal clinical practice.

In case of suspected ocular flare-up, the ophthalmologist may consider performing a full or partial ophthalmological work-up based on clinical need. The clinical-instrumental data obtained from the ophthalmological assessments will be collected in a standardised electronic database according to the variables described in the case report form (CRF).

ELIGIBILITY:
Inclusion Criteria:

* For GCA group:

  * Patients older than 18 years with clinically suspected or confirmed gigantocellular arteritis.
  * Newly found visual involvement with suspected or confirmed correlation with vasculitis.
  * Ability to express valid consent to study enrolment.
* For control group:

  * Patients older than 18 years with the ability to express valid consent to study enrolment.
  * Newly diagnosed acute visual impairment with GCA phenotypes (e.g. AION, CRAO) but without any correlation with vasculitis aetiology.

Exclusion Criteria:

* Pre-existing ophthalmological pathologies that may modify best visual acuity and/or alter ophthalmological semeiotics.
* Concomitant active viral, bacterial, fungal and parasitic infections, including active or latent tuberculosis treated for less than 4 weeks and HIV, hepatitis C virus (HCV)

  /hepatitis B virus (HBV) infections, involving the eyes and orbital cavities.
* Concomitant systemic inflammations not attributable to GCA (inflammatory diseases in treatment-free remission are not excluded).
* Any other condition judged by the investigators to be a contraindication of eligibility

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive adult patients presenting with transient or permanent visual impairment, with or without associated vasculitic pathology, at the emergency department or ophthalmology outpatient clinic.
Sampling Method: Non-Probability Sample
Enrollment: 762 (Estimated)
Dates: Start 2024-06-27 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Comparison of specific signs in A-AION vs. NA-AION and GCA-related CRAO vs. non-GCA-related. | Since beginning of study for 6 years
  The primary outcome is a comparison of the frequency of the various semeiological findings by multi-parametric evaluation (visual field, fundus oculi, OCT, OCT-A, FAG, ICGA), among the main pathological ocular alterations of arteritic and non-arteritic aetiology, such as A-AION Vs. NA-AION and CRAO from arteritis Vs. CRAO from other causes.

SECONDARY OUTCOMES:
Frequency of the pathological phenotypes of GCA visual involvement | Since beginning of study for 6 years
  A description of the prevalence of the GCA visual phenotypes, including the potential co-existence of several of them, for example, paracellular retinal ischemia as in PAMM, choroidal and papillary ischemia).
Correlating the various clinical findings with different ophthalmological methods for each GCA ocular phenotype, at baseline. | At subject's enrollment
  Integration of clinical findings at baseline with ophthalmological methods such as visual acuity, campimetry, FAG, ICGA, OCT, and OCT-A in various pathological visual conditions.
Correlating the various clinical findings with different ophthalmological methods for each GCA ocular phenotype, during follow-up | Since patient's enrollment for 6 months
  Integration of clinical findings during follow-up with ophthalmological methods such as visual acuity, campimetry, FAG, ICGA, OCT, and OCT-A in various pathological visual conditions.
Visual impairment evolution over time, analysing predictors of improved or worsened evolution. | Since patient's enrollment for 6 months
  Temporal evolution of the visual acuity and semeiological findings after therapy and correlation with prognosis.

OTHER OUTCOMES:
Identification of GCA biohumoral markers correlated with specific GCA ocular phenotypes | Since beginning of study for 6 years
Identification of GCA biohumoral markers correlated with visual prognosis | Since beginning of study for 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Invernizzi, Prof., Principal Investigator — ASST Fatebenefratelli Sacco
Locations (1):
- ASST Fatebenefratelli-Sacco, Milan, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: Undecided